CLINICAL TRIAL: NCT03671395
Title: The DCU Running Injury Surveillance Centre (RISC) Study: A Prospective Investigation of Factors Relating to Running Injuries
Brief Title: The DCU Running Injury Surveillance Centre Study: A Prospective Investigation of Factors Relating to Running Injuries
Acronym: DCU RISC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dublin City University (Other)
Collaborators: Insight Centre for Data Analytics (Other)
Responsible Party: Sponsor
Other Study IDs: SFI12/RC/2289
Record Dates: First submitted 2018-05-02; First posted 2018-09-14 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Musculoskeletal Injury
Keywords: Running Injuries; Motion Analysis; Biomechanics; Inertial Measurement Unit; Sensor Technology; Kinetic; Kinematic; Injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to prospectively investigate the relationship between a number of clinical and biomechanical variables and running-related injuries among a group of novice and recreational runners over a two year time period. To date, the incidence of running injuries among runners is high, with a lack of prospective research investigating the factors related to injury. It is thought that loading in excess of the tissues capabilities may be be a contributing factor to sustaining a running related injury. As such, this study hypothesizes that biomechanical factors may be related to injury.

Healthy participants will perform a battery of clinical tests at baseline, as well as completing a survey that details their injury history and training habits. Kinematic and kinetic motion analysis will be used as participants perform a series of functional movements and a treadmill run. Enrolled participants will be monitored for the occurrence of running-related injuries via email for the duration of the study.

DETAILED DESCRIPTION:
Recruitment:

Novice and recreational runners will be recruited via emails, posters and social media. A novice runner is defined as a person who has not been running on a regular basis during the last year and completed ≤10km total training volume per week during the preceding year. A recreational runner will be defined as a person who runs a minimum of 10km per week, for at least six months prior to inclusion in the study.

Study Protocol:

Upon screening for inclusion and exclusion, participants will complete a baseline evaluation. This will consist of 1.) A survey, 2.) A battery of clinical tests and 3.) Motion analysis testing. A description of each component is detailed below.

1. Survey:

   This survey will be self-reported by each participant. The aim of this survey is to detail each participants history of injuries and training habits. Questions are deigned based on previous survey designs relating to running injuries.
2. Battery of clinical tests:

   The battery of physical performance tests will include: The foot posture index, the navicular drop, goniometry of the hip and ankle, dynamometry of the hip abductors, hip extensors, knee extensors, knee flexors and plantar flexors.
3. Motion analysis testing:

This will be broken into two components; a functional movement protocol and a treadmill run. During these components, motion will be tracked using wearable inertial sensors (Shimmer, Dublin, Ireland) and two forceplates (AMTI, Watertown, MA, USA). A 17-camera 3D motion analysis system (Vicon, Oxford, United Kingdom) will capture data at a sampling rate of 200 Hz. Reflective markers will be applied to the skin using specific anatomical landmarks to map their location. The functional movement protocol will consist of a series of jumping and landing movements, including double leg and single leg counter movement jumps, unilateral hopping, single leg drop landings and single leg drop jumps. Following this, participants will complete a run to fatigue. Motion analysis data will be captured at the end and start of this run. Fatigue will be determined by a reported rate of perceived exertion score of 17 (very hard) on the BORG Scale and a heart rate of 85% of the heart rate max, as determined by the Karvonen Formula (220-age).

Participants will then resume their normal training regime. Participants will be tracked for injuries via email over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Runners aged 18-65
* Run minimum once per week

Exclusion Criteria:

* No lower limb injury within the last three months

An injury will be defined as:

* Any muscle, bone, tendon or ligament pain in the lower back, hip, groin, thigh, leg, knee, foot, ankle and toe that caused the participant to stop or restrict their running.
* The pain must last for at least 7 days or 3 consecutive scheduled training sessions, or require the participant to consult a physician or other health care professional.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Novice and recreation runners.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
The occurrence of a running-related injury | 6 week intervals from enrollment in the study, up to the total study time period of 2 years.
  Participants will be followed up on a 6 week basis via email. A running-related injury will be defined as any muscle, bone, tendon or ligament pain in the lower back, hip, groin, thigh, leg, knee, foot, ankle and toe that caused the participant to stop or restrict their running. The pain must last for at least 7 days or 3 consecutive scheduled training sessions, or require the participant to consult a physician or other health care professional.
Peak loading (N/s) during running and jumping movements. | One two hour session on day one of enrollment into the study.
  This data will be derived from the inertial measurement units (Shimmer, Dublin, Ireland) attached to the legs and pelvis and using forceplate data (AMTI, Watertown, USA).
Rate of loading (N/s2) during running. | One two hour session on day one of enrollment into the study
  This data will be derived from the inertial measurement units (Shimmer, Dublin, Ireland) attached to the legs and pelvis and using forceplate data (AMTI, Watertown, USA).

SECONDARY OUTCOMES:
Peak range of motion (degrees) at the knee, hip and ankle during running. | During a 15 minute run during one two hour session on day 1 of enrollment into the study.
  Captured and extracted via Vicon Motion Analysis Software (Oxford, UK).
Injury history in the past 2 years. | 10 minute questionnaire on day one of enrollment into the study.
  Frequency, type and severity measured via online survey.
Training history- type | 10 minute questionnaire on day one of enrollment into the study.
  Typical type of training (Distance, interval, hill, speed), measured via online survey.
Training history-frequency | 10 minute questionnaire on day one of enrollment into the study.
  Typical frequency (sessions per week) measured via online survey.
Training history- mileage | 10 minute questionnaire on day one of enrollment into the study.
  Typical mileage (km/week) and duration (minutes/session) measured via online survey.
Training history- duration | 10 minute questionnaire on day one of enrollment into the study.
  Typical session duration (minutes/session) measured via online survey.

OTHER OUTCOMES:
Foot Posture Index (Scale, scoring from -12 to +12) | Measured during a single two hour session on day one of enrollment into the study.
  Measure of static foot position.
Navicular drop (mm) | Measured during a single two hour session on day one of enrollment into the study.
  Measure of dynamic foot pronation.
Hip internal and external rotation range (degrees) | One two hour session on day one of enrollment into the study.
  Measured in sitting using a clinometer mobile application.
Hip extension range (degrees) | Measured during a single two hour session on day one of enrollment into the study.
  Measured using the modified Thomas Test.
Knee to wall test (degrees) | Measured during a single two hour session on day one of enrollment into the study.
  Measured using a clinometer mobile application.
Isometric muscle strength of the hip abductors bilaterally (N/kg). | Measured during single two hour session on day one of enrollment into the study.
  Measured bilaterally in the supine position via hand held dynamometer (J-Tech Limited).
Isometric muscle strength of the hip extensors bilaterally (N/kg). | Measured during single two hour session on day one of enrollment into the study.
  Measured bilaterally in the prone position via hand held dynamometer (J-Tech Limited).
Isometric muscle strength of the knee extensors bilaterally (N/kg). | Measured during single two hour session on day one of enrollment into the study.
  Measured bilaterally in a seated position via hand held dynamometer using a fixation belt(J-Tech Limited).
Isometric muscle strength of the knee flexors bilaterally (N/kg). | Measured during single two hour session on day one of enrollment into the study.
  Measured bilaterally in a seated position via hand held dynamometer using a fixation belt (J-Tech Limited).
Isometric muscle strength of the plantar flexors bilaterally (N/kg). | Measured during single two hour session on day one of enrollment into the study.
  Measured in a prone position via hand held dynamometer using a fixation belt (J-Tech Limited).

CONTACTS AND LOCATIONS:
Overall Officials: Aoife Burke, Principal Investigator — Dublin City University, Insight Centre for Data Analytics; Sarah Dillon, Principal Investigator — Dublin City University, Insight Centre for Data Analytics; Dr Kieran Moran, Principal Investigator — Dublin City University, Insight Centre for Data Analytics
Locations (1):
- Dublin City University, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data may be shared to allow future analysis by other researchers.

REFERENCES:
- [Background] Bredeweg SW, Kluitenberg B, Bessem B, Buist I. Differences in kinetic variables between injured and noninjured novice runners: a prospective cohort study. J Sci Med Sport. 2013 May;16(3):205-10. doi: 10.1016/j.jsams.2012.08.002. Epub 2012 Aug 24. PMID 22921763
- [Background] Buist I, Bredeweg SW, Lemmink KA, van Mechelen W, Diercks RL. Predictors of running-related injuries in novice runners enrolled in a systematic training program: a prospective cohort study. Am J Sports Med. 2010 Feb;38(2):273-80. doi: 10.1177/0363546509347985. Epub 2009 Dec 4. PMID 19966104
- [Background] Ghani Zadeh Hesar N, Van Ginckel A, Cools A, Peersman W, Roosen P, De Clercq D, Witvrouw E. A prospective study on gait-related intrinsic risk factors for lower leg overuse injuries. Br J Sports Med. 2009 Dec;43(13):1057-61. doi: 10.1136/bjsm.2008.055723. Epub 2009 Feb 18. PMID 19228665
- [Background] Hespanhol Junior LC, Pena Costa LO, Lopes AD. Previous injuries and some training characteristics predict running-related injuries in recreational runners: a prospective cohort study. J Physiother. 2013 Dec;59(4):263-9. doi: 10.1016/S1836-9553(13)70203-0. PMID 24287220
- [Background] Lun V, Meeuwisse WH, Stergiou P, Stefanyshyn D. Relation between running injury and static lower limb alignment in recreational runners. Br J Sports Med. 2004 Oct;38(5):576-80. doi: 10.1136/bjsm.2003.005488. PMID 15388542
- [Background] Malisoux L, Nielsen RO, Urhausen A, Theisen D. A step towards understanding the mechanisms of running-related injuries. J Sci Med Sport. 2015 Sep;18(5):523-8. doi: 10.1016/j.jsams.2014.07.014. Epub 2014 Aug 12. PMID 25174773
- [Background] Nielsen RO, Buist I, Parner ET, Nohr EA, Sorensen H, Lind M, Rasmussen S. Predictors of Running-Related Injuries Among 930 Novice Runners: A 1-Year Prospective Follow-up Study. Orthop J Sports Med. 2013 May 2;1(1):2325967113487316. doi: 10.1177/2325967113487316. eCollection 2013 Jan-Jun. PMID 26535228